CLINICAL TRIAL: NCT06615310
Title: The Relationship of Ultrasonographic Parameters Used in the Evaluation of Dysphagia in Stroke Patients With Swallowing Severity
Brief Title: Ultrasonographic Parameters in Stroke Patients With Dysphagia
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Cansin Medin, associate proffesor, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: 2024-41
Record Dates: First submitted 2024-09-13; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Dysphagia
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dysphagia: 3 Points and above according to the EAT-10 scale
  Interventions: Other: ultrasonograpic evaluotion
- non-dysphagia: Under 3 points on the EAT-10 scale
  Interventions: Other: ultrasonograpic evaluotion

INTERVENTIONS:
Other: ultrasonograpic evaluotion — The distance between the hyoid and thyroid cartilage, the volume of the geniohyoid, digastric anterior, sternohyoid and thyrohyoid muscles will be evaluated by ultrasound.

SUMMARY:
ultrasonographic parameters in stroke patients with dysphagia

ELIGIBILITY:
Inclusion Criteria: Diagnosis of stroke,

* Agreeing to participate in the study,
* Cognitive competence to understand the test instructions
* Communication skills to respond to the test instructions.

Exclusion Criteria:

* Presence of a neurological disease other than stroke that will cause difficulty in swallowing, -Being illiterate,
* refusing to participate in the study,
* jaw joint problem,
* surgical intervention in the neck area that will affect ultrasound measurements,
* infected open wound

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been diagnosed with stroke at Istanbul Physical Therapy and Rehabilitation Training and Research Hospital and enrolled in a rehabilitation program will be divided into 2 groups according to the presence of dysphagia (3 points and above according to the EAT-10 scale).
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
muscle volume of thyrohyoid | baseline
  the thickness of the muscle will be measured by ultrasound

SECONDARY OUTCOMES:
muscle volume of sternohyoid | baseline
  the thickness of the muscle will be measured by ultrasound

IPD SHARING:
Plan to Share IPD: Undecided